CLINICAL TRIAL: NCT00180648
Title: Plasma Determination of Glucagon-like Peptide 2 as a Predictor of Recovery in Adults With Acute Intestinal Failure
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Centre for Ocular Research & Education, Canada (Other); St Mark's Hospital Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 04/Q0405/83
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2008-05

CONDITIONS: Short Bowel Syndrome
Keywords: Short Bowel Syndrome; Intestinal Failure; Glucagon Like Peptide 2; Parenteral Nutrition
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure; Hyperphagia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the theory that the plasma level of Glucagon like peptide 2 (GLP-2) in patients with intestinal failure can predict their clinical recovery.

DETAILED DESCRIPTION:
When major segments of small bowel have been removed surgically, or damaged by disease, the length of the residual bowel may be inadequate to maintain overall nutrition and the net result is described as "intestinal failure".

Without medical intervention, patients with intestinal failure become malnourished and dehydrated because their remaining intestine is unable to absorb enough water, vitamins and other nutrients from the ingested food. Intravenous feeding offers life saving treatment but causes complications like infections and liver problems. It also poses enormous strain on day to day life.

Glucagon like peptide 2 (GLP-2) is a naturally occurring hormone (or chemical messenger) that is able to increase the surface area of the intestinal lining (or mucosal mass) and the absorptive efficiency of the remaining intestine.

Intestinal failure patients in whom not only parts of the small bowel but also the large bowel have had to be surgically removed have been shown to have a markedly impaired rise in GLP-2 levels following meals, in contrast to patients with a preserved large bowel who have increased levels of GLP-2 and are known to have much better functional adaptation.

From this we hypothesise that the GLP-2 level is directly related to, and could predict, clinical recovery in intestinal failure as measured by Amount of parenteral nutrition required Length of hospital stay Mortality

We also aim to compare GLP-2 levels of patients with acute intestinal failure with that of patients with chronic intestinal failure as well as healthy controls

ELIGIBILITY:
Inclusion Criteria:

* Men and woman, aged 18 years of age or older at the time of signing the informed consent form.
* Referral to or direct admission to St. Mark's Hospital.
* Acute intestinal failure resulting in TPN dependency as a result of major intestinal resection performed during admission to St. Mark's or at the referring hospital.

Exclusion Criteria:

* Inability to give consent or comply with the study.
* Inability to take test meal (unable to be tested)
* Severe renal impairment (interference with GLP-2 excretion)
* Severe uncorrected anaemia (preventing additional blood-letting)
* Uncontrolled diabetes mellitus (risk of hyperglycaemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Intestinal failure patients at St Mark's hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Forbes, Principal Investigator — University College London Hospitals

REFERENCES:
- See also: Web site devoted to the study of the glucagon-like peptides — http://www.glucagon.com